CLINICAL TRIAL: NCT02672956
Title: Comparison of Different Umbilical Port Entry Techniques in Terms of Cosmetic Results
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zeynep Kamil Maternity and Pediatric Research and Training Hospital (Other)
Responsible Party: Principal Investigator, Mehmet Baki Senturk, Principal investigator, Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 129
Record Dates: First submitted 2016-01-21; First posted 2016-02-03 (Estimated); Last update posted 2022-03-29 (Actual); Status verified 2022-03

CONDITIONS: Cicatrix
MeSH Terms: conditions — Cicatrix | interventions — Surgical Instruments

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Supraumbilical entry group (Experimental): Umbilical port will be insert to supra umbilical area.
  Interventions: Procedure: Ten mm trocar
- Intraumbilical entry group (Experimental): Umbilical port will be insert to intra umbilical area.
  Interventions: Procedure: Ten mm trocar
- Infraumbilical group (Experimental): Umbilical port will be insert to infra umbilical area.
  Interventions: Procedure: Ten mm trocar

INTERVENTIONS:
Procedure: Ten mm trocar

SUMMARY:
Investigators selected participants who operated by laparoscopic technique due to any gynecologic indication according to random number table. The ten mm trocar was inserted supraumbilical, infraumbilical and intraumbilical. The verres needle was not used in all of patients. One month after we evaluated umbilical scar by used vancouver scar scale and compared results of vancouver scar scale.

ELIGIBILITY:
Inclusion Criteria:

* Participant with eligible for laparoscopic surgery

Exclusion Criteria:

* Participant with umbilical scar due to previous surgery, burn eg.

Ages: 20 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 105 (Actual)
Dates: Start 2015-09 (Actual); Primary Completion 2017-09 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
The results of vancouver scar scale | One month

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet Baki Şentürk, MD, Principal Investigator — Zeynep Kamil Maternity and Pediatric Research and Training Hospital
Locations (1):
- Zeynep Kamil Maternity and Pediatric Research and Training Hospital, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Background] Kim E, Kim D, Lee S, Lee H. Minimal-scar laparoscopic adjustable gastric banding (LAGB). Obes Surg. 2009 Apr;19(4):500-3. doi: 10.1007/s11695-008-9713-6. Epub 2008 Oct 7. PMID 18839082
- [Result] Park SK, Olweny EO, Best SL, Tracy CR, Mir SA, Cadeddu JA. Patient-reported body image and cosmesis outcomes following kidney surgery: comparison of laparoendoscopic single-site, laparoscopic, and open surgery. Eur Urol. 2011 Nov;60(5):1097-104. doi: 10.1016/j.eururo.2011.08.007. Epub 2011 Aug 12. PMID 21856076
- [Result] Nozaki T, Ichimatsu K, Watanabe A, Komiya A, Fuse H. Longitudinal incision of the umbilicus for laparoendoscopic single site adrenalectomy: a particular intraumbilical technique. Surg Laparosc Endosc Percutan Tech. 2010 Dec;20(6):e185-8. doi: 10.1097/SLE.0b013e3181f70a2a. PMID 21150398
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/21856076
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Longitudinal+Incision+of+the+Umbilicus+for+Laparoendoscopic+Single+Site+Adrenalectomy%3A+A+Particular+Intraumbilical+Technique
- See also: Related Info — http://www.ncbi.nlm.nih.gov/pubmed/?term=Minimal-Scar+Laparoscopic+Adjustable+Gastric+Banding+(LAGB)